CLINICAL TRIAL: NCT05305950
Title: Exploring Barriers and Facilitators to Mitigate Disparities in Access to OT/PT in Pediatric Cancer Survivors
Brief Title: Barriers and Facilitators in Access to OT/PT in Pediatric Cancer Survivors
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0893; NCI-2021-12740 (Other: NCI-CTRP Clinical Trials Reporting Process)
Record Dates: First submitted 2022-03-09; First posted 2022-03-31 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare administrators: Healthcare administrators at MD Anderson Cancer Center and the sister institutions
  Interventions: Other: Patient population
- Physicians/referring providers: Physicians/referring providers and the occupational therapy (OT) and physical therapy (PT) therapists at MD Anderson Cancer Center and the sister institutions
  Interventions: Other: Patient population

INTERVENTIONS:
Other: Patient population — Questionnaire, standard of care

SUMMARY:
This study aims to identify the modifiable facilitators and barriers to occupational and physical therapy care for children during and after cancer treatment that may be contributing to disparities in health outcomes. The investigators will identify these facilitators and barriers by surveying and interviewing healthcare administrators at MD Anderson Cancer center. The investigators will also survey and interview physicians, advanced practice providers, and occupational and physical therapists to obtain their feedback on these issues.

ELIGIBILITY:
Aim 1 Inclusion Criteria:

* Employed as an administrator at MD Anderson Cancer Center and the sister institutions and working in the areas of pediatrics, survivorship, cancer control, health policy, and rehabilitation services.

Aim 2 Inclusion Criteria:

* Employed as a referring provider (e.g., oncologist, surgeon, advanced care practitioner), or an OT/PT therapist at MD Anderson Cancer Center and the sister institutions.

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify modifiable barriers to occupational and physical therapy care for children during cancer treatment that may be contributing to disparities in health outcomes. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karen Moody, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org